

A series of randomised controlled N-of-1 trials in patients who have discontinued or are considering discontinuing statin use due to muscle-related symptoms to assess if atorvastatin treatment causes more muscle symptoms than placebo

**Informed Consent Form** 

PROTOCOL NUMBER: ISRCTN30952488

## **Appendix 7 StatinWISE Informed Consent Form**



## Name of Principal Investigator:

| 1. Patient Initials | 2. Patient Screening ID | 3. Site ID |
|---------------------|-------------------------|------------|

| Statement | | | Please initial<br>each box |
|---|---|---|---|
| I confirm that I have read the information sheet d<br>study and given a copy to keep. I have had the op<br>and have these answered satisfactorily. | | | |
| I understand that my participation is voluntary an giving any reason, and without my medical care o | | | |
| I understand that relevant sections of my medical looked at by individuals from the sponsor of the tand responsible persons authorised by the sponsor the NHS Trust, where it is relevant to my taking paindividuals to have access to my records. | rial (London School of Hygiene & Tropical Moor, from ethics and regulatory authorities, or | edicine)<br>from | |
| I understand that my personal details will be kept<br>be available to LSHTM Clinical Trial Unit staff to po | | | |
| I understand that the information collected about<br>used to support other research in the future, and<br>used in future ethically approved research project | | | |
| I give permission for a copy of this consent form, available to the LSHTM Clinical trials Unit. | | | |
| I agree to take part in the StatinWISE study. | | | |
| Printed name of participant | Signature of participant | Date | |
| confirm that I have explained the study informatio<br>participant and that he/sl | n accurately to, and was understood to the l<br>he has freely given their consent to participa | | knowledge by, the |
| Printed name of person obtaining consent | Signature of person obtaining consent | Date | Date |

1 copy of participant, 1 for investigator file and 1 for medical notes.